CLINICAL TRIAL: NCT05641337
Title: Research on Optimal Strategy of Hypoglycemic Therapy for Cirrhosis With Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, xiaolong zhao, Chief Physician, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-10-cirrhosis with DM
Record Dates: First submitted 2022-11-06; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Liver Cirrhosis; Diabetes
Keywords: Liver cirrhosis; diabetes; time in range; insulin intensive therapy; new combination therapy
MeSH Terms: conditions — Liver Cirrhosis; Diabetes Mellitus | interventions — insulin degludec, insulin aspart drug combination; Metformin; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group with new combination therapy (Experimental): The hypoglycemic scheme of the experimental group was that the initial dose of Insulin Degludec and Insulin Aspart was 0.3U/kg multiplied by the patient's weight, plus 5 mg of linagliptin and 0.5 g of metformin three times a day.
  Interventions: Drug: Insulin Degludec and Insulin Aspart
- group with intensive insulin therapy (Active Comparator): group was treated with intensive insulin therapy.The initial total amount of insulin is 0.5U/kg, of which 40% is basal insulin and 20% is aspart insulin before three meals
  Interventions: Drug: Insulin Degludec and Insulin Aspart

INTERVENTIONS:
Drug: Insulin Degludec and Insulin Aspart — The hypoglycemic scheme of the experimental group was that the initial dose of Insulin Degludec and Insulin Aspart was 0.3U/kg multiplied by the patient's weight, plus 5 mg of linagliptin and 0.5 g of metformin three times a day. The control group was treated with traditional four needle insulin.
  Other Names: metformin; linagliptin

SUMMARY:
Poor blood glucose control in liver cirrhosis can aggravate the poor prognosis of patients. Under the background of the increasing number of liver cirrhosis patients with metabolic abnormalities, how to optimize treatment is particularly important. The traditional treatment of diabetes at the stage of liver cirrhosis is limited to insulin intensive therapy, but the incidence of hypoglycemia is high, blood sugar fluctuates greatly, and multiple injections are required. Research shows that insulin therapy has an increased overall mortality compared with non insulin therapy. We used metformin,Ryzodeg and an oral DDP IV enzyme inhibitor as the core combination according to the special pathological mechanism of elevated blood glucose in liver cirrhosis . After preliminary experiments, we found that the program was stable and was not easy to have hypoglycemia, and there was no traditional risk of lactic acid poisoning caused by metformin. We designed an open randomized controlled clinical study, Compared with the traditional insulin intensive treatment scheme, this new combination scheme was compared whether it could improve the blood glucose level, the incidence of hypoglycemia and lactic acid level, the incidence of cirrhosis complications, and the long-term survival rate of liver disease. This study is helpful to optimize the hypoglycemic treatment of cirrhosis with diabetes, and improve the blood glucose and long-term prognosis, The positive evidence of this study contributes to the consensus or guidelines for the treatment of cirrhosis with diabetes.

DETAILED DESCRIPTION:
Cirrhosis with diabetes refers to the increase of blood sugar in cirrhosis, including cirrhosis before or after diabetes. It has a special pathophysiological mechanism that liver factors participate in blood glucose regulation. Poor blood glucose control in liver cirrhosis can aggravate the poor prognosis of patients. Under the background of the increasing number of liver cirrhosis patients with metabolic abnormalities, how to optimize treatment is particularly important. The traditional treatment of diabetes at the stage of liver cirrhosis is limited to insulin intensive therapy, but the incidence of hypoglycemia is high, blood sugar fluctuates greatly, and multiple injections are required. Research shows that insulin therapy has an increased overall mortality compared with non insulin therapy. We used metformin, ,Ryzodeg and an oral DDP IV enzyme inhibitor as the core combination according to the special pathological mechanism of elevated blood glucose in liver cirrhosis from multiple links. After preliminary experiments, we found that the program was stable and was not easy to have hypoglycemia, and there was no traditional risk of lactic acid poisoning caused by metformin. We designed an open randomized controlled clinical study, Compared with the traditional insulin intensive treatment scheme, this new combination scheme was compared whether it could improve the blood glucose level, the incidence of hypoglycemia and lactic acid level, the incidence of cirrhosis complications, and the long-term survival rate of liver disease. This study is helpful to optimize the hypoglycemic treatment of cirrhosis with diabetes, and improve the blood glucose and long-term prognosis of such patients, The positive evidence of this study contributes to the consensus or guidelines for the treatment of cirrhosis with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Age 18-70 years
* Patients with elevated blood sugar who meet the diabetes standard or have been treated with hypoglycemic drugs
* random finger or venous serum blood glucose more than 14 mmol/L

Exclusion Criteria:

* Those unwilling to participate or unable to cooperate;
* Child-pugh score is greater than 12;
* Glomerular filtration rate<60ml/min/1.73m2;
* Patients with cardiac insufficiency;
* Patients with asymptomatic hypoglycemia;
* Pregnant patients were excluded;
* Patients with advanced liver cancer;
* Blood pressure is less than 90/60mmHg;
* Chronic liver disease plus acute or subacute liver failure;
* Patients with drug induced blood glucose disorder, such as glucocorticoids, contraceptives, etc;
* fingertip oxygen saturation less than 95% without oxygen inhalation;
* Autoimmune liver cirrhosis is currently taking hormone.
* Type 1 diabetes.
* Pancreatogenic diabetes, such as primary hemochromatosis, hepatolenticular degeneration, alcoholic pancreatitis, autoimmune diseases involving the pancreas, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
time in range | two weeks
  time in range
Blood lactic acid level | two week
  Blood lactic acid level
Compound adverse events | two week
  includetimes of hypolgycemia attack，severe hypoglycemia attack and serum lactic acid more than 2.2 mmol/L, complications of liver cirrhosis within two week

SECONDARY OUTCOMES:
mean blood glucose | two weeks
  mean blood glucose
Time above range | two weeks
  Time above range
Time below range | two weeks
  Time below range
Blood lactic acid | two weeks
  Blood lactic acid
Glycated Albumin | two week
  Glycated Albumin
three month mortality | three months
  three month mortality
Six month mortality | six months
  Six month mortality
Incidence rate of complications of liver cirrhosis within three months | three months
  Incidence rate of complications of liver cirrhosis within three months
Incidence rate of complications of liver cirrhosis within six months | six months
  Incidence rate of complications of liver cirrhosis within six months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Zhao, PhD, Study Chair — Shanghai Public Health Clinical Center
Locations (1):
- Xiaolong Zhao, Shanghai, Shanghai Municipality, China